CLINICAL TRIAL: NCT02132897
Title: Fed Bioequivalence Study of Carbamazepine Controlled Release Formulations in Healthy Male Uruguayan Subjects
Brief Title: Fed Bioequivalence Study of CBZ Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Clinical Pharmacology Research Bdbeq S.A. (Other)
Responsible Party: Principal Investigator, Francisco E. Estevez-Carrizo, M.D., Chief Medical Officer, Center for Clinical Pharmacology Research Bdbeq S.A.
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: BDBEQ-CBZ400/EUFUY-023
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Bio-equivalence Study; Fed Conditions
Keywords: Antiepileptic; Carbamazepine; Bio-equivalence; Fed; Crossover
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Carbamazepine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TR (Test - Reference) (Other): Sequence : Auration CR 400 Single Dose/Tegretol CR 400 Single Dose
  Interventions: Drug: Auration CR Tablets 400 Single Dose-Tegretol CR 400 Single Dose
- RT (Reference - Test) (Other): Sequence: Tegretol CR 400 Single Dose/Auration CR 400 Single Dose
  Interventions: Drug: Tegretol CR 400 Single Dose-Auration CR 400 Single Dose

INTERVENTIONS:
Drug: Auration CR Tablets 400 Single Dose-Tegretol CR 400 Single Dose — Carbamazepine CR Tablets 400 milligrams is given orally with 250 mL of water at room temperature.
  Other Names: Carbamazepine; Carbamazepine CR; Carbamazepine CR 400 millligrams
  Arms: TR (Test - Reference)
Drug: Tegretol CR 400 Single Dose-Auration CR 400 Single Dose — Auration CR 400 milligrams Single Dose is given orally with 250 mL of water at room temperature.
  Other Names: Carbamazepine; Carbamazepine CR; Carbamazepine CR 400
  Arms: RT (Reference - Test)

SUMMARY:
Controlled release Carbamazepine (CBZ) is a antiepileptic, antineuralgic and mood stabilizer drug. The CR formulation of CBZ is slowly absorbed and the elimination half life varies with time due to metabolism autoinduction.

The primary objective of this study is to estimate the bioequivalence of the new brand generic product (Auration(R) CR) 400 mg manufactured in Uruguay vs. the innovative product (Tegretol(R) CR) 400 mg manufactured in Brasil, under fed conditions. The secondary objective will be evaluation of safety issues.

The study design will be randomized two sequences, two periods and crossover. For a power of not less than 80% sample size was estimated to be 20 healthy male subjects. Products will be administered with food (high calories/high fat breakfast) after an overnight fast.

Time vs. concentration curves will be built for each subject and formulation and Area Under Curve (AUC0240) will be estimated using the trapezoid rule, the AUC 0-inf. (from time 0 to infinity) will be estimated using the formula Cz/Ke, Cmax will be taken from the individual curves.

This parameters will be statistically processed with the WinNonlin 6.3 Pharmacokinetics/Statistic software in order to prove bioequivalence between the study products.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or smokers of less than 5 cigarettes/day, within the age range of 18 to 50 years.
* Body Mass Index (BMI = weight/height2) greater than or equal to 18.5 kg/m2 and less than or equal to 24.9 kg/m2.
* No clinically significant findings in the physical examination, 12-lead electrocardiogram (ECG) and vital signs (blood pressure between 100-140/58-90 mmHg, heart rate between 50-99 beats/min, temperature between 35.8ºC and 37.6ºC, respiration rate between 12 and 20 breaths/minute)
* No clinical laboratory values outside of the acceptable range as per protocol, unless the Principal Investigator or Sub-investigator decides that they are not clinically significant (NCS).
* Availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements.
* The subject agrees to abstain from alcohol, coffee and other food and drinks containing methylxanthines (mate, tea, cola, chocolate) for 48hours, and grapefruit containing food and beverages for 72 hours prior study drug administration and during each study period.

Exclusion Criteria:

* Known history of hypersensitivity to Carbamazepine and/or related drugs.
* Positive test for hepatitis B surface antigen, hepatitis C or HIV.
* Known history of gastrointestinal (e.g: gastritis, inflammatory bowel disease, celiac disease), cardiac, pulmonary, endocrine, musculoskeletal, neurological, hematological, immunological, hepatic or renal disease, or malignancies, unless deemed NCS by the Principal Investigator or Sub-investigator.
* Any history of peptic ulcer disease or gastrointestinal (GI) bleeding.
* Any history of gastrointestinal surgery (except for appendectomy).
* Presence of any significant physical or organ abnormality.
* Any illness during the 4 weeks before this study, unless deemed NCS by the Clinical Investigator or Sub-investigator.
* Any history or evidence of psychiatric or psychological disease, unless deemed NCS by the Clinical Investigator or Sub-investigator.
* Any history of asthma (after 12 years of age).
* Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens).
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Any history of drug and psychoactive medicines abuse.
* Any recent history of alcohol abuse (less than 1 year).
* Use of any prescription medication within 14 days preceding this study.
* Use of vaccinations within 30 days preceding this study.
* Use of over-the-counter (OTC) medication within the 7 days preceding this study (except for spermicidal/barrier contraceptive products, sunscreen and sunblock products).
* Participation as a plasma donor in a plasmapheresis program within 7 days preceding this study.
* Blood donations within 60 days preceding and after this study.
* Participation in a clinical trial with an investigational drug within 180 days preceding this study, and agreement not to participate in a clinical trial for 180 days after this study.
* Intolerance to venipuncture.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AUC0-240 | 10 days
  Area Under the CBZ Concentration vs. time curve from sample time point 0 hour to sample time point 240 hour.
AUC0-inf | 0 to 240 hours
  Area Under the CBZ Concentrations vs, time curve from sample time point 0 hour to sample time point 240 hours plus extrapolation to infinity of the terminal concentration slope.
Cmax | 12 to 48 hours
  The maximum concentration in the CBZ concentrations vs. time curves for each subject and each formulation.

SECONDARY OUTCOMES:
AE | 31 days
  Recording of all adverse events (AE) occurring during the study: expected, unexpected and serious (SAE) from tree different sources. The AEs may be clinical occurrences, abnormal labs or ECG alterations.

OTHER OUTCOMES:
Tmax | 12 to 48 hours
  Time from 0 concentration sample point to the Cmax sample point.
Ke | From 48 to 240 hours
  The constant rate of elimination (Ke) is the slope of the terminal phase of the CBZ concentration vs. time curve.
T1/2e | 48 to 240 hours
  It is the time that CBZ concentration, in the elimination (terminal) phase, fall off by half.
Vital signs | 20 days
  Measuring of blood pressure, heart rate, body temperature and ventilation rate.
Admission and discharge screening | 21 days
  Laboratory analysis and ECG performed prior to admission to the clinic and prior to discharge from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco E. Estevez-Carrizo, M.D., Study Director — Center for Clinical Pharmacology Research Bdbeq S.A.; Francisco T. Estevez-Parrillo, M.D., Principal Investigator — Center for Clinical Pharmacology Research Bdbeq S.A.
Locations (1):
- Center for Clinical Pharmacology Research Bdbeq S.A. Italian Hospital, Montevideo, Montevideo Department, Uruguay